CLINICAL TRIAL: NCT01610804
Title: Choroidal Thickness Measurements During CSCR Treatment Applying EDI-OCT Technology
Brief Title: Choroidal Thickness Measurements During Central Serous Chorioretinopathy (CSCR) Treatment
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Caroline Brandl, MD, University Hospital Regensburg
Other Study IDs: CSCR2011
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Choroidal Thickness

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CSCR-Patients: Patients suffering from Central Serous Chorioretinopathy
- Healthy Subjects: Healthy subjects with (assumed) normal choroidal thickness

SUMMARY:
The purpose of this study is to determine changes in choroidal thickness in patients with Central Serous Chorioretinopathy (CSCR) during the first 3 months after initial diagnosis via Enhanced-Depth-Imaging-Spectral-Domain-Optical-Coherence-Tomography (EDI-OCT).

Study hypothesis: Since exudative changes in the choroid seem to constitute the primary pathology of CSCR, changes in choroidal thickness compared to healthy eyes should be present and be visible using EDI-OCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial diagnosis of CSCR and no treatment so far

Exclusion Criteria:

* Therapy (drugs/laser) due to CSCR

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with reduction of vision due to Central Serous Chorioretinopathy
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Gamulescu, PD Dr. med., Study Chair — University Hospital Regensburg
Locations (1):
- University Hospital Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Imamura Y, Fujiwara T, Margolis R, Spaide RF. Enhanced depth imaging optical coherence tomography of the choroid in central serous chorioretinopathy. Retina. 2009 Nov-Dec;29(10):1469-73. doi: 10.1097/IAE.0b013e3181be0a83. PMID 19898183
- [Background] Margolis R, Spaide RF. A pilot study of enhanced depth imaging optical coherence tomography of the choroid in normal eyes. Am J Ophthalmol. 2009 May;147(5):811-5. doi: 10.1016/j.ajo.2008.12.008. Epub 2009 Feb 20. PMID 19232559